CLINICAL TRIAL: NCT01881178
Title: The Effect of a Nutritional Supplement Product Containing Cactus Fruit Juice (Nopalea) on C-Reactive Protein (NOPALEA)
Brief Title: The Effect of a Nutritional Supplement Product Containing Cactus Fruit Juice (Nopalea) on C-Reactive Protein
Acronym: NOPALEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Mattie (Other)
Responsible Party: Sponsor-Investigator, Mark Mattie, Associate Professor, University of Bridgeport
Organization: University of Bridgeport (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nopalea
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2013-06

CONDITIONS: Inflammation
Keywords: CRP; Nopalea; Fruit; Juice
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apricot (Active Comparator): Supplement: Apricot Juice
  Interventions: Dietary Supplement: NOPALEA
- Nopalea (Experimental): Supplement: Nopalea
  Interventions: Dietary Supplement: NOPALEA

INTERVENTIONS:
Dietary Supplement: NOPALEA

SUMMARY:
This study has been developed to investigate the anti-inflammatory effects of a commercial product (Nopalea) containing Prickly Pear Cactus Fruit Juice in healthy adults. The research method employs a double blind, placebo controlled, and time-series (repeat measures) design with high-sensitivity C-Reactive Protein (HS-CRP) serving as a marker for inflammation - testing for levels of CRP at time points: baseline (pre-test), 8 weeks (60 days) and 12 weeks (90 days). The final time point (i.e., 12 weeks) will serve as the post-test. It is expected that baseline CRP levels in healthy participants will decline.

ELIGIBILITY:
Live within traveling distance of the research center. Access to a telephone in their residence. Between 35 and 75 years of age Not currently ingesting Nopalea Not pregnant, planning to become pregnant, or nursing a child Not currently taking anti-inflammatory medications Medically stable - i.e. no recent major change in the last 3 weeks of prescription or non- prescription medication Not diagnosed with Type 1 Diabetes Not diagnosed with depression Not diagnosed with an acquired or congenital immune system deficiency

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
HS-CRP | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark e Mattie, Study Director — UBCNM
Locations (1):
- Trivita Wellness Center, Scottsdale, Arizona, United States